CLINICAL TRIAL: NCT05178095
Title: Artificial Intelligence in Colonic Polyp Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Hedenström, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dnr 2020-01951
Record Dates: First submitted 2021-11-15; First posted 2022-01-05 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Polyp of Colon; Adenoma Colon; Gastrointestinal Neoplasms
Keywords: colonoscopy; artificial intelligence
MeSH Terms: conditions — Colonic Polyps; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI (Experimental): Colonoscopy with AI
  Interventions: Device: Artificial intelligence
- No AI (Placebo Comparator): Colonoscopy without AI
  Interventions: Device: No Artificial Intelligence

INTERVENTIONS:
Device: Artificial intelligence — Colonoscopy with the aid of artificial intelligence for the detection of colonic polyps
  Arms: AI
Device: No Artificial Intelligence — Colonoscopy without the aid of artificial intelligence for the detection of colonic polyps
  Arms: No AI

SUMMARY:
A randomized, controlled study investigating the potential benefits of artificial intelligence (AI) in the detection of colonic polyps during outpatient colonoscopy. Randomization between the use of AI and no AI is performed before the study procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients without IBD referred for colonoscopy

Exclusion Criteria:

* Age < 40 years
* Not willing to participate

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
ADR | 1 hour
  Adenoma detection rate

SECONDARY OUTCOMES:
APC | 1 hour
  Adenomas per colonoscopy
Procedural time | 1 hour
  The number of minutes required to complete the colonoscopy withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Björn Lindkvist, Study Director — Sahlgrenska University Hospital
Locations (1):
- Dr Per Hedenström, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scholer J, Alavanja M, de Lange T, Yamamoto S, Hedenstrom P, Varkey J. Impact of AI-aided colonoscopy in clinical practice: a prospective randomised controlled trial. BMJ Open Gastroenterol. 2024 Jan 30;11(1):e001247. doi: 10.1136/bmjgast-2023-001247. PMID 38290758